CLINICAL TRIAL: NCT03003325
Title: The Benefit/Risk Profile of Pegylated Proline-Interferon Alpha-2b (AOP2014) Added to the Best Available Strategy Based on Phlebotomies in Low-risk Patients With Polycythemia Vera (PV). The Low-PV Randomized Trial
Brief Title: The Benefit/Risk Profile of AOP2014 in Low-risk Patients With PV
Acronym: Low-PV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: FROM- Fondazione per la Ricerca Ospedale di Bergamo- ETS (Other)
Collaborators: AOP Orphan Pharmaceuticals AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Low-PV
Record Dates: First submitted 2016-11-03; First posted 2016-12-28 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Polycythemia Vera
Keywords: low risk of thrombosis; Interferon
MeSH Terms: conditions — Polycythemia Vera | interventions — Blood Specimen Collection; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phlebotomies + ASA (Active Comparator): Conventional treatment based on phlebotomies and low dose (100 mg) of acetylsalicylic acid (ASA)
  Interventions: Procedure: Phlebotomies; Drug: ASA
- Phlebotomies + ASA + AOP2014 (Experimental): Conventional treatment based on phlebotomies, low dose (100 mg) of acetylsalicylic acid (ASA) plus the addition of 100 µg of Pegylated Proline-Interferon alpha-2b (AOP2014) once every 14 days (subcutaneously).
  Interventions: Drug: AOP2014; Procedure: Phlebotomies; Drug: ASA

INTERVENTIONS:
Drug: AOP2014 — AOP2014 will be supplied to the patients as pre-filled auto-injection pens, containing 250 µg of active drug (0.5 ml solution for injection). One pen may be used twice within a time period of 4 weeks. Hence investigators will provide one prefilled pen at every monthly visit. AOP2014 will be self-injected subcutaneously by patients once every 14 days at the single doses of 100 µg (0.2 ml).
  Other Names: Pegylated-Proline-Interferon α-2b, P1101
  Arms: Phlebotomies + ASA + AOP2014
Procedure: Phlebotomies — According to current common clinical practice the regimen must be selected accordingly to maintain the recommended level of HCT< 45%. Once normalization of the hematocrit has been achieved, blood counts at regular intervals (every 4 weeks) will establish the frequency of future phlebotomies. Sufficient blood should be removed to maintain the hematocrit below 45%.
  Other Names: blood removing
Drug: ASA — 100 mg/daily of ASA is recommended (when there are not contraindications) according with current guidelines for this risk class of patients
  Other Names: Acetylsalicylic Acid

SUMMARY:
The Low-PV study is a multicenter, phase II, randomized trial aimed to assess whether the addition of Pegylated Proline-interferon-alpha-2b to the best therapeutic current strategy available based on phlebotomies and low dose acetylsalicylic acid (ASA) could improve the efficacy of treatment of patients with PV at low risk of thrombosis (younger than 60 years and without prior vascular events), in term of control of recommended level of hematocrit < 45%, over a period of 12 months.

DETAILED DESCRIPTION:
It is an independent, investigator-generated, pragmatic trial including adult PV patients (aged 18-60) diagnosed according to World Health Organization 2008 criteria within the last 3 years before inclusion, without history of thrombosis and younger than 60 years ('low risk' patients).

Eligible patients are randomized to be treated with the best available therapy (recommended for this risk class, standard arm) based on phlebotomy including administration of low-dose (100 mg/daily) of acetylsalicylic acid (ASA, when there are not contraindications) OR Pegylated Proline-Interferon alpha-2b (AOP2014) every 2 weeks in addition to the recommended available regimen (experimental arm), for up to 12 months. The allocation of patients to study arms is 1:1 and stratification at randomization will be performed according to age category (< 50 years old or > 50 years old) and time from diagnosis (naϊve or non-naϊve). Naive patients are defined as new cases coming to observation, diagnosed for the first time just before study entry and never treated; non-naive patients are old cases (diagnosis not older than 3 years before study entry) undergoing therapy with phlebotomy and/or low doses of ASA.

Primary endpoint (PEp) is defined by the proportion (%) of patients who maintain the median value of hematocrit (HCT) below 45% during 12 months of treatment in each arm, without progression of disease and no need of any extra-protocol cytoreductive drug (responder patients).

Secondary endpoints include evaluation of hematological and molecular response, histological remission and safety profile of the protocol therapy.

Before randomization all patients undergo phlebotomies in order to reach an HCT below 45%.

After randomization, according to current common clinical practice the regimen of phlebotomies must be selected accordingly to maintain the recommended level of HCT< 45%. Once normalization of the HCT has been achieved, blood counts at regular intervals (every 4 weeks) will establish the frequency of future phlebotomies. Sufficient blood is recommended to be removed in order maintain the hematocrit below 45%. Supplemental iron therapy should not be administered.

All patients receive low-dose of ASA (100 mg/daily) as recommended by the current guidelines for low-risk subjects with PV.

Patients allocated in the experimental group receive in addition a pre-filled auto-injection pen for the subcutaneous auto-administration (into the abdominal skin or the thigh) of 100 µg of Pegylated Proline-Interferon alpha-2b (AOP2014) once every 14 days.

Patient visits are scheduled every month (4 weeks) for 12 months to assess and perform a reliable calculation of the primary end-point (% of patients with median HCT levels <45%).

At each monthly visit a pre-filled auto-injection pen is delivered to the patients who have been randomized in the experimental arm.

Assuming an expected drop-out rate of 12%, a total sample size of 150 patients (75 randomized in each group) will be randomized to reject the null hypothesis that the proportion of patients achieving the primary endpoint is 50% in favor of the alternative hypothesis that this proportion is 75% when AOP2014 is added to the phlebotomy based- therapy, with a power of 80% and an alpha error of 0.05 (two-tailed).

Two interim-analysis are planned when 50 and 100 of randomized patients have completed the 12 months study, respectively, in order to evaluate and supervise both safety and primary endpoint. The Lan and DeMets (1983) spending function with O'Brien-Fleming type boundaries will be employed to preserve the overall two-sided type I error rate for effectiveness at the 0.05 level, regardless of the timing of the analysis.

The results of the second interim analysis carried out at in April 2020 indicated a significant higher efficacy of the experimental arm than standard arm. The composite primary end-point was reached in 84% in patients of Ropeginterferon arm vs. 60% in standard arm (p=0.008, Odds Ratio=3.5, 95% CI: 1.3-10.4). This result, according to the statistical evaluation for futility and efficacy, reveals that , the null hypothesis is already been proven with first 100 patients randomized and cannot change in the future when 150 patients will enter the study. Therefore the data safety monitoring board and the steering committee agree that the accrual of new patients can be interrupted with 127 patients included.

The primary endpoint assessment is performed after the completion of the first 12 months of therapy for all subjects enrolled ('core study').

A period of 12 months is expected for completion of the enrolment / randomization phase. The 'core study' itself will take 12 months of treatment per patient.

Based on results from the 'core study' the extension phase will continue as follows:

1. After 12 month patients who meet the primary endpoint following either conventional or experimental therapy will enter the extension phase and remain on their current regimen.
2. non-responders, not meeting the primary endpoint after 12 months of conventional therapy will be switched to the experimental treatment.
3. non-responder, not meeting the primary endpoint after 12 months of experimental therapy will be switched to conventional treatment.

This extension phase will last for another 12 months from the Last Visit Last Patient included (LVLP) into the core study (matching cases 1 and 2 as defined above). Based on this, the overall length of the study is expected to cover a period of 36 months from the First Patient Included (FPI).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years
* Diagnosis of Polycythemia Vera according to World Health Organization 2016 criteria
* Diagnosis of Polycythemia Vera including a recent bone marrow (BM) biopsy (performed within 3 years prior randomization in the study) and never treated with cytoreductive drugs
* HCT<45%
* Ability and willingness to comply with all study requirements
* Signed written informed consent.

Exclusion Criteria:

* Any previous well documented cardiovascular PV-related events (see Appendix 1 for description)
* Previous cytoreductive drugs
* Known hypersensitivity or contraindications to the Investigational Medicinal Product (Pegylated Proline-Interferon alpha-2b) including:

evidence of severe retinopathy (e.g. cytomegalovirus retinitis, macular degeneration) or clinically relevant ophthalmological disorder (due to diabetes mellitus or hypertension); thyroid dysfunction not adequately controlled; patients tested positively with Thyroglobulin antibody and / or TPOAb at screening; documented autoimmune disease at screening or in the medical history; history or presence of depression requiring treatment with antidepressant; any risk of suicide at screening or previous suicide attempts;

* Previous exposure to a non-pegylated or pegylated interferon α
* Clinically relevant pulmonary infiltrates, pneumonia, and pneumonitis
* Systemic infections, e.g. hepatitis B, hepatitis C, or HIV at screening
* Significant liver (AST or alanine aminotransferase > 2.5 times ULN) or renal disease (creatinine > 2 mg/ml)
* Presence of any life-threatening condition or of any disease (e.g. cancer) that is likely to significantly shorten life expectancy
* History of active substance or alcohol abuse within the last year
* Any condition that in the opinion of the investigator would jeopardize the evaluation of efficacy or safety or be associated with poor adherence to the protocol
* Pregnant or lactating women and women*/men of childbearing potential who are not using or are not willing to use any effective means of contraception (i.e. sexual abstinence, hormonal contraceptive, intra-uterine device, barrier method such as diaphragms or condoms, surgical methods).

  * Pregnancy test will be performed in order to ascertain negativity of human chorionic gonadotropin (β-hCG) test and confirm that childbearing women are not pregnant.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 127 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Number of patients who maintains the median value of HCT< 45%, along 12 months, on number of patients randomized in each arm, per cent | 12 months
  For each patient the median value of HCT percentage will be calculated from all measurements detected and reported every month (from baseline to 12-month visit or study end). A patient will be defined as responder (achieving PEp) when he maintains the median value of HCT < 45%, after undergoing treatments according to this protocol, for up 12 months.
  A patient will be defined as non-responder (not achieving PEp) when
  1. Does not maintain the median value of HCT < 45%, after undergoing treatments according to this protocol, for up 12 months, or
  2. Is in need of any additional chemotherapeutic and/or cytoreductive treatment aimed to manage disease due to disease progression.

SECONDARY OUTCOMES:
Median number of phlebotomies performed | 12 months, 24 months
  1. The total number of phlebotomies will be calculated for each patients during 12 months of therapy (and then 24 months);
  2. Based on values obtained from point (1) in each arm-group of patients, the median number of phlebotomies performed in each therapy group will be calculated (and compared) after 12 and 24 months of therapy (or completion of the study)
Number of patients achieving hematological response (as defined below in 'Description') on number of patients randomized in each arm, per cent, | 12 months, 24 months
  For each patient the median value of HCT (%), absolute white blood cells (WBCs) count and absolute platelets (PLTs) count will be calculated from all measurements detected and reported at least every month (from baseline to 12-month visit and then to 24-month visit/study completion). A patient will be defined as achieving hematological response when the median values of HCT < 45%, WBCs count < 10 x10*9/L and PLTs count < 400 x10*9/L is observed after 12 months of therapy (or 24 months). The proportion of patients who maintains this response after 24 months (or study completion) will be calculated (and compared) in each arm.
Proportion (rate per cent) of patients with not palpable spleen | 12 months, 24 months
  The proportion (rate per cent) of patients with not palpable spleen will be calculated in each arm as the ratio of number of patients with resolution of splenomegaly or persistence of not palpable spleen at palpation with respect to baseline, on number of patients randomized in each arm, after 12 and 24 months (study completion) of therapy, per cent.
Janus kinase-2 allele burden reduction or complete molecular remission | 12 months, 24 months
  Quantitative Janus kinase-2 measurements (central lab facility) will be performed at baseline and after 12 months of therapy for all patients; Janus kinase-2 assessment will be performed also after 24 months for patients receiving interferon (experimental therapy). Reduction of allele burden in each patient (with respect to baseline) will be assessed according to Jovanovic et al, Leukemia 2013.
  The proportion (rate per cent) of patients with Janus kinase-2 allele burden reduction or remission will be calculated in each arm (and compared).
Bone marrow histological remission | 24 months
  Defined as presence of age-adjusted normocellularity and disappearance of trilinear hyperplasia, and absence of >grade 1 reticulin fibrosis. It will be assessed in each patient and then the proportion (rate per cent) of patients with bone marrow histological remission will be calculated in each arm (and compared).
Incidence and frequence of thrombotic and hemorrhagic events occurred | 12 months, 24 months
  The number of events will be recorded any time during the study in order to assess the frequency ,every 12 months and at completion of the study, and their incidence in each arm and whole population. Comparison between arms will be performed.
Number of adverse events occurred | 12 months, 24 months
  Incidence, causality and intensity of clinical relevant adverse events will be assessed in each arm and compared all over the study.
  The rate of assigned treatment withdrawal due to any protocol drug-related toxicity occurred any time will be compared. Number of adverse events, expressed as frequency in each arm, will be calculated (as ratio of number of patient experiencing adverse on the the number of patients randomized in each arm) and compared

OTHER OUTCOMES:
Quality of Life (QoL) | 12 months, 24 months
  Impact of PV and therapy on subjects will be evaluated through assessment of symptoms burden using Functional Assessment of cancer Therapy-Anaemia (FACT-An) and Myeloproliferative Neoplasm Symptom Assessment Form total symptom score (MPN-SAF TSS) questionnaires, that will be administered to subjects trimonthly

CONTACTS AND LOCATIONS:
Overall Officials: Tiziano Barbui, Professor, Study Chair — Fondazione per la Ricerca Ospedale Maggiore di Bergamo (FROM)
Locations (23):
- Italy (23):
  - U.O. Ematologia, Ospedale Casa Sollievo della Sofferenza Istituto di Ricovero e Cura a Carattere Scientifico, San Giovanni Rotondo, (FG) Puglia
  - U.O. Ematologia con Trapianto, Azienda Universitaria Ospedaliera Consorziale - Policlinico Bari, Bari, Apulia
  - Azienda Ospedaliera Universitaria Federico II di Napoli, Napoli, Campania
  - Divisione Ematologia Policlinico S. Orsola - Malpighi, Bologna, Emilia-Romagna
  - Clinica Ematologica, Azienda Ospedaliero-Universitaria "Santa Maria della Misericordia", Udine, Friuli Venezia Giulia
  - UCSC Ematologia, Fondazione Policlinico Universitario "Agostino Gemelli"Università Cattolica del Sacro Cuore, Rome, Lazio
  - UOC Ematologia, ASST Papa Giovanni XXIII, Bergamo, Lombardy
  - Divisione Oncoematologia, Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - Divisione Ematologia ASST, Grande Ospedale Metropolitano Niguarda, Milan, Lombardy
  - Divisione Ematologia, ASST di MONZA - Ospedale San Gerardo di Monza, Monza, Lombardy
  - Divisione Ematologia, Fondazione IRCCS Policlinico San Matteo, Pavia, Lombardy
  - U.O. Ematologia, Ospedale di Circolo e Fondazione Macchi Varese, Varese, Lombardy
  - S.C. Ematologia Azienda Ospedaliera S. Croce e Carle Cuneo, Cuneo, Piedmont
  - SCDU Ematologia, A.O.U. Maggiore della Carità, Novara, Piedmont
  - S.C. Ematologia, AOU- Presidio Ospedaliero Molinette, Turin, Piedmont
  - Unità Operativa Complessa di Emostasi Azienda Ospedaliero-Universitario "Policlinico Vittorio-Emanuele - Presidio Ospedaliero Ferrarotto, Catania, Sicily
  - UOC Ematologia, Azienda Ospedaliera Universitaria Policlinico "G. Martino", Messina, Sicily
  - Divisione Ematologia Azienda Ospedaliera Universitaria Policlinico "Paolo Giaccone" Palermo, Palermo, Sicily
  - SOD Ematologia AUOC Azienda Ospedaliero-Universitaria "Careggi", Florence, Tuscany
  - Clinica Medica I Azienda Ospedaliera di Padova, Padua, Veneto
  - Divisione Ematologia, Ospedale Borgo Roma, Verona, Veneto
  - Divisione Ematologia, Ospedale San Bortolo, Vicenza, Veneto
  - IRCCS Ospedale San Raffaele, Milan

IPD SHARING:
Plan to Share IPD: No
No plan has been defined yet about sharing of IPD

REFERENCES:
- [Background] Kralovics R, Passamonti F, Buser AS, Teo SS, Tiedt R, Passweg JR, Tichelli A, Cazzola M, Skoda RC. A gain-of-function mutation of JAK2 in myeloproliferative disorders. N Engl J Med. 2005 Apr 28;352(17):1779-90. doi: 10.1056/NEJMoa051113. PMID 15858187
- [Background] Scott LM, Tong W, Levine RL, Scott MA, Beer PA, Stratton MR, Futreal PA, Erber WN, McMullin MF, Harrison CN, Warren AJ, Gilliland DG, Lodish HF, Green AR. JAK2 exon 12 mutations in polycythemia vera and idiopathic erythrocytosis. N Engl J Med. 2007 Feb 1;356(5):459-68. doi: 10.1056/NEJMoa065202. PMID 17267906
- [Background] Passamonti F, Elena C, Schnittger S, Skoda RC, Green AR, Girodon F, Kiladjian JJ, McMullin MF, Ruggeri M, Besses C, Vannucchi AM, Lippert E, Gisslinger H, Rumi E, Lehmann T, Ortmann CA, Pietra D, Pascutto C, Haferlach T, Cazzola M. Molecular and clinical features of the myeloproliferative neoplasm associated with JAK2 exon 12 mutations. Blood. 2011 Mar 10;117(10):2813-6. doi: 10.1182/blood-2010-11-316810. Epub 2011 Jan 11. PMID 21224469
- [Background] Vannucchi AM, Rotunno G, Bartalucci N, Raugei G, Carrai V, Balliu M, Mannarelli C, Pacilli A, Calabresi L, Fjerza R, Pieri L, Bosi A, Manfredini R, Guglielmelli P. Calreticulin mutation-specific immunostaining in myeloproliferative neoplasms: pathogenetic insight and diagnostic value. Leukemia. 2014 Sep;28(9):1811-8. doi: 10.1038/leu.2014.100. Epub 2014 Mar 12. PMID 24618731
- [Background] Barbui T, Barosi G, Birgegard G, Cervantes F, Finazzi G, Griesshammer M, Harrison C, Hasselbalch HC, Hehlmann R, Hoffman R, Kiladjian JJ, Kroger N, Mesa R, McMullin MF, Pardanani A, Passamonti F, Vannucchi AM, Reiter A, Silver RT, Verstovsek S, Tefferi A; European LeukemiaNet. Philadelphia-negative classical myeloproliferative neoplasms: critical concepts and management recommendations from European LeukemiaNet. J Clin Oncol. 2011 Feb 20;29(6):761-70. doi: 10.1200/JCO.2010.31.8436. Epub 2011 Jan 4. PMID 21205761
- [Background] Najean Y, Rain JD. The very long-term evolution of polycythemia vera: an analysis of 318 patients initially treated by phlebotomy or 32P between 1969 and 1981. Semin Hematol. 1997 Jan;34(1):6-16. No abstract available. PMID 9025157
- [Background] Treatment of polycythaemia vera by radiophosphorus or busulphan: a randomized trial. "Leukemia and Hematosarcoma" Cooperative Group, European Organization for Research on Treatment of Cancer (E.O.R.T.C.). Br J Cancer. 1981 Jul;44(1):75-80. doi: 10.1038/bjc.1981.150. PMID 7020738
- [Background] Marchioli R, Finazzi G, Landolfi R, Kutti J, Gisslinger H, Patrono C, Marilus R, Villegas A, Tognoni G, Barbui T. Vascular and neoplastic risk in a large cohort of patients with polycythemia vera. J Clin Oncol. 2005 Apr 1;23(10):2224-32. doi: 10.1200/JCO.2005.07.062. Epub 2005 Feb 14. PMID 15710945
- [Background] Barosi G, Vannucchi AM, De Stefano V, Pane F, Passamonti F, Rambaldi A, Saglio G, Barbui T, Tura S. Identifying and addressing unmet clinical needs in Ph-neg classical myeloproliferative neoplasms: a consensus-based SIE, SIES, GITMO position paper. Leuk Res. 2014 Feb;38(2):155-60. doi: 10.1016/j.leukres.2013.09.008. Epub 2013 Sep 19. PMID 24378116
- [Background] Barosi G, Mesa R, Finazzi G, Harrison C, Kiladjian JJ, Lengfelder E, McMullin MF, Passamonti F, Vannucchi AM, Besses C, Gisslinger H, Samuelsson J, Verstovsek S, Hoffman R, Pardanani A, Cervantes F, Tefferi A, Barbui T. Revised response criteria for polycythemia vera and essential thrombocythemia: an ELN and IWG-MRT consensus project. Blood. 2013 Jun 6;121(23):4778-81. doi: 10.1182/blood-2013-01-478891. Epub 2013 Apr 16. PMID 23591792
- [Background] Marchioli R, Finazzi G, Specchia G, Cacciola R, Cavazzina R, Cilloni D, De Stefano V, Elli E, Iurlo A, Latagliata R, Lunghi F, Lunghi M, Marfisi RM, Musto P, Masciulli A, Musolino C, Cascavilla N, Quarta G, Randi ML, Rapezzi D, Ruggeri M, Rumi E, Scortechini AR, Santini S, Scarano M, Siragusa S, Spadea A, Tieghi A, Angelucci E, Visani G, Vannucchi AM, Barbui T; CYTO-PV Collaborative Group. Cardiovascular events and intensity of treatment in polycythemia vera. N Engl J Med. 2013 Jan 3;368(1):22-33. doi: 10.1056/NEJMoa1208500. Epub 2012 Dec 8. PMID 23216616
- [Background] Gisslinger H, Ludwig H, Linkesch W, Chott A, Fritz E, Radaszkiewicz T. Long-term interferon therapy for thrombocytosis in myeloproliferative diseases. Lancet. 1989 Mar 25;1(8639):634-7. doi: 10.1016/s0140-6736(89)92142-9. PMID 2564458
- [Background] Tefferi A, Hudgens S, Mesa R, Gale RP, Verstovsek S, Passamonti F, Cervantes F, Rivera C, Tencer T, Khan ZM. Use of the Functional Assessment of Cancer Therapy--anemia in persons with myeloproliferative neoplasm-associated myelofibrosis and anemia. Clin Ther. 2014 Apr 1;36(4):560-6. doi: 10.1016/j.clinthera.2014.02.016. Epub 2014 Mar 14. PMID 24636526
- [Background] Emanuel RM, Dueck AC, Geyer HL, Kiladjian JJ, Slot S, Zweegman S, te Boekhorst PA, Commandeur S, Schouten HC, Sackmann F, Kerguelen Fuentes A, Hernandez-Maraver D, Pahl HL, Griesshammer M, Stegelmann F, Doehner K, Lehmann T, Bonatz K, Reiter A, Boyer F, Etienne G, Ianotto JC, Ranta D, Roy L, Cahn JY, Harrison CN, Radia D, Muxi P, Maldonado N, Besses C, Cervantes F, Johansson PL, Barbui T, Barosi G, Vannucchi AM, Passamonti F, Andreasson B, Ferrari ML, Rambaldi A, Samuelsson J, Birgegard G, Tefferi A, Mesa RA. Myeloproliferative neoplasm (MPN) symptom assessment form total symptom score: prospective international assessment of an abbreviated symptom burden scoring system among patients with MPNs. J Clin Oncol. 2012 Nov 20;30(33):4098-103. doi: 10.1200/JCO.2012.42.3863. Epub 2012 Oct 15. PMID 23071245
- [Background] Barbui T, Carobbio A, Rambaldi A, Finazzi G. Perspectives on thrombosis in essential thrombocythemia and polycythemia vera: is leukocytosis a causative factor? Blood. 2009 Jul 23;114(4):759-63. doi: 10.1182/blood-2009-02-206797. Epub 2009 Apr 16. PMID 19372254
- [Background] Kiladjian JJ, Mesa RA, Hoffman R. The renaissance of interferon therapy for the treatment of myeloid malignancies. Blood. 2011 May 5;117(18):4706-15. doi: 10.1182/blood-2010-08-258772. Epub 2011 Mar 9. PMID 21389325
- [Background] Kiladjian JJ, Cassinat B, Chevret S, Turlure P, Cambier N, Roussel M, Bellucci S, Grandchamp B, Chomienne C, Fenaux P. Pegylated interferon-alfa-2a induces complete hematologic and molecular responses with low toxicity in polycythemia vera. Blood. 2008 Oct 15;112(8):3065-72. doi: 10.1182/blood-2008-03-143537. Epub 2008 Jul 23. PMID 18650451
- [Background] Quintas-Cardama A, Abdel-Wahab O, Manshouri T, Kilpivaara O, Cortes J, Roupie AL, Zhang SJ, Harris D, Estrov Z, Kantarjian H, Levine RL, Verstovsek S. Molecular analysis of patients with polycythemia vera or essential thrombocythemia receiving pegylated interferon alpha-2a. Blood. 2013 Aug 8;122(6):893-901. doi: 10.1182/blood-2012-07-442012. Epub 2013 Jun 19. PMID 23782935
- [Background] Jovanovic JV, Ivey A, Vannucchi AM, Lippert E, Oppliger Leibundgut E, Cassinat B, Pallisgaard N, Maroc N, Hermouet S, Nickless G, Guglielmelli P, van der Reijden BA, Jansen JH, Alpermann T, Schnittger S, Bench A, Tobal K, Wilkins B, Cuthill K, McLornan D, Yeoman K, Akiki S, Bryon J, Jeffries S, Jones A, Percy MJ, Schwemmers S, Gruender A, Kelley TW, Reading S, Pancrazzi A, McMullin MF, Pahl HL, Cross NC, Harrison CN, Prchal JT, Chomienne C, Kiladjian JJ, Barbui T, Grimwade D. Establishing optimal quantitative-polymerase chain reaction assays for routine diagnosis and tracking of minimal residual disease in JAK2-V617F-associated myeloproliferative neoplasms: a joint European LeukemiaNet/MPN&MPNr-EuroNet (COST action BM0902) study. Leukemia. 2013 Oct;27(10):2032-9. doi: 10.1038/leu.2013.219. Epub 2013 Jul 17. PMID 23860450
- [Derived] Barbui T, Vannucchi AM, De Stefano V, Carobbio A, Ghirardi A, Carioli G, Masciulli A, Rossi E, Ciceri F, Bonifacio M, Iurlo A, Palandri F, Benevolo G, Pane F, Ricco A, Carli G, Caramella M, Rapezzi D, Musolino C, Siragusa S, Rumi E, Patriarca A, Cascavilla N, Mora B, Cacciola E, Mannarelli C, Loscocco GG, Guglielmelli P, Gesullo F, Betti S, Lunghi F, Scaffidi L, Bucelli C, Vianelli N, Bellini M, Finazzi MC, Tognoni G, Rambaldi A. Ropeginterferon versus Standard Therapy for Low-Risk Patients with Polycythemia Vera. NEJM Evid. 2023 Jun;2(6):EVIDoa2200335. doi: 10.1056/EVIDoa2200335. Epub 2023 May 15. PMID 38320126
- [Derived] Barbui T, Vannucchi AM, De Stefano V, Masciulli A, Carobbio A, Ferrari A, Ghirardi A, Rossi E, Ciceri F, Bonifacio M, Iurlo A, Palandri F, Benevolo G, Pane F, Ricco A, Carli G, Caramella M, Rapezzi D, Musolino C, Siragusa S, Rumi E, Patriarca A, Cascavilla N, Mora B, Cacciola E, Mannarelli C, Loscocco GG, Guglielmelli P, Betti S, Lunghi F, Scaffidi L, Bucelli C, Vianelli N, Bellini M, Finazzi MC, Tognoni G, Rambaldi A. Ropeginterferon alfa-2b versus phlebotomy in low-risk patients with polycythaemia vera (Low-PV study): a multicentre, randomised phase 2 trial. Lancet Haematol. 2021 Mar;8(3):e175-e184. doi: 10.1016/S2352-3026(20)30373-2. Epub 2021 Jan 18. PMID 33476571
- [Derived] Kiladjian JJ, Barbui T. From leeches to interferon: should cytoreduction be prescribed for all patients with polycythemia vera? Leukemia. 2020 Nov;34(11):2837-2839. doi: 10.1038/s41375-020-0984-9. Epub 2020 Jul 16. No abstract available. PMID 32678292